CLINICAL TRIAL: NCT01403181
Title: Effect of Boceprevir Therapy on HCV-specific T Cell Responses: Perspectives of Immune Monitoring and Immune Therapy
Brief Title: Effect of Boceprevir on HCV-specific T Cell Responses
Acronym: Boce-Par
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Carlo Ferrari, MD, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: AZOSPA
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; T cells; cytokines; cytotoxicity; proliferation
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera and peripheral blood lymphomononuclear cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic hepatitis C: * 10 naïve genotype 1 chronic hepatitis C patients treated with PEG plus RBV (control arm)
  * 20 naïve genotype 1 chronic hepatitis C patients treated with a response guided therapy consisting of Boceprevir in combination with PEG plus RBV (experimental arm)
  Interventions: Drug: Boceprevir

INTERVENTIONS:
Drug: Boceprevir — In the experimental arm boceprevir (800 mg orally three times daily), PEG-IFN and ribavirin will be given for 24 weeks after the lead-in; the patients who will have undetectable HCV-RNA at week 8 will stop treatment at week 28; those who will be HCV-RNA positive at any visit between week 8 and 24 will receive an additional 20 weeks of PEG + RBV. Treatment will be discontinued if HCV-RNA is positive at week 24.
  Immunological analysis will be performed longitudinally at the following time points: week -4, 0, 4 (end of lead-in), 8, 12, 24, 48, week 24 of follow-up. HCV-RNA will be quantified at the same time points and viremia will be correlated with immunological data.
  Other Names: Peginterferon alfa-2b and ribavirin

SUMMARY:
Analysis of HCV-specific T cell responses in patients treated with boceprevir to assess whether therapy can induce restoration of the T cell function and to what extent this recovery can be achieved

DETAILED DESCRIPTION:
Reconstitution of the antiviral T cell function may represent a component of the anti-viral effect of protease inhibitors. If T cell responsiveness is restored under therapy, potentiation of anti-viral T cell functions by exogenous T cell stimulation might be exploited to complement and to further improve response to available therapies. Monitoring the T cell function might also be useful to predict more accurately response to therapy.

To address these issues, phenotype and function of HCV-specific T cells will be analyzed longitudinally before, during and after therapy in naïve genotype 1 chronic hepatitis C patients treated with peginterferon plus ribavirin or with peginterferon and ribavirin plus boceprevir. To analyze the global CD4 and CD8 reactivity against all structural and non-structural HCV proteins a wide panel of peptides corresponding to the whole HCV genome of genotype 1 will be employed. To further analyze CD8 reactivity, HLA-A2/peptide tetramers will be used in HLA-A2 positive patients to directly quantify ex vivo HCV-specific CD8 cells circulating in the peripheral blood.The T cell function will be analyzed as capacity of expansion in vitro, cytokine production and cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Male or female, aged from 18 to 70 years old, inclusive.
* Willing and able to provide written informed consent
* Chronic HCV infection for at least 6 month prior to baseline (Day 1) in subjects currently positive for HCV-RNA and anti-HCV antibody documented by:
* A positive anti-HCV antibody test, positive HCV-RNA assay, or HCV genotype test at least 6 month prior to baseline (Day 1) or
* A liver biopsy performed prior to baseline (Day 1) with evidence of chronic HCV infection
* Subjects must have liver biopsy results (performed no more than two years prior the screening) indicating the absence of cirrhosis
* HCV infection limited to genotype 1
* Detectable plasma HCV-RNA at screening
* BMI between 18 and 36 Kg/m2
* Eligible subjects must also be HCV treatment-naïve, defined as no prior exposure to PEG-INF and ribavirin, and must be eligible to standard of care therapy with PEG/RBV
* Subjects must have the following laboratory parameters at screening:

ALT and AST ≤ 5 x upper limit of normal range (ULN) Hemoglobin (Hb) ≥ 12 g/dl WBC ≥ 2.500 cells/μL with absolute neutrophil count ≥ 1500 cells/μL If a woman of childbearing potential, must have negative serum β-human chorionic gonadotropin (β-HCG) pregnancy test documented at the screening visit and a negative serum or urine pregnancy test before the first dose of study drug to ensure that they are not pregnant at the time of starting treatment A female subjects of childbearing potential and nonvasectomized male subjects with a female partners of childbearing potential must agree that they and their partner will use effective contraception (two separate forms of contraception simultaneously, one of which must be a male condom with spermicide) from screening throughout the duration of study treatment and for at least 7 months

Exclusion Criteria:

* Pregnant women or women who may wish to become pregnant during the course of the study
* Male with a female who is pregnant or is planning to become pregnant within seven month the study of anticipated last dose of ribavirin
* Evidence of infection or co-infection with a no-genotype 1 HCV-strain
* History of hemoglobinopathy
* History of sarcoidosis
* History of invasive malignancy diagnosed or treated within 5 years.
* Untreated or significant psychiatric illnesses including severe depression, schizophrenia, psychosis, history of a suicide attempt
* Co-infection with HBV or HIV
* Chronic use of systemic immunosuppressive agents
* Presence of autoimmune disorders; subjects with treated hypothyroidism with normal TSH may be enrolled
* History of significant cardiac disease
* Clinical evidence of chronic pulmonary disease
* Known cirrhosis
* History of solid organ transplantation
* Suspicion of hepatocellular carcinoma
* Chronic liver disease of a non-HCV etiology
* Ongoing alcohol abuse
* History of clinical relevant drug abuse
* Positive urine screen for cocaine, opiate etc, or methadone use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Naïve genotype 1 chronic hepatitis C patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Levels of HCV-specific T cell functions before, during and after therapy to measure functional restoration induced by therapy | 2 years
  Capacity of expansion, cytokine production (IFN-γ, IL-2 and TNF-α) and cytotoxicity expressed by HCV-specific T cells will be analyzed longitudinally at different time points before, during and after therapy

SECONDARY OUTCOMES:
Correlation of quality and intensity of pre-treatment HCV-specific T cell responses with outcome of therapy | 2 years
  To assess whether different levels of efficiency of pre-treatment antiviral T cell responses can predict response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ferrari, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Unit of Infectious Diseases and Hepatology, Parma, Italy, Italy